CLINICAL TRIAL: NCT06849193
Title: Dynamic Prediction Model for Patients with Unresectable Biliary Malignancies Receiving Systemic Chemotherapy Combined with Immunotherapy: a Multicenter, Observational Study
Acronym: BTCICTY-001
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Third Affiliated Hospital of Soochow University (Other); Jiangsu Cancer Institute & Hospital (Other); The First Affiliated Hospital, University of Science and Technology of China (Other); Zhejiang Cancer Hospital (Other); Shanghai Zhongshan Hospital (Other); Yunnan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Director of interventional and Vascular Surgery Department, Zhongda Hospital
Other Study IDs: 2024040196
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Unresectable Biliary Tract Cancer; Dynamic Prediction Model; Immunotherapy
Keywords: Unresectable Biliary Tract Cancer; immunotherapy; Dynamic prediction model; systemic chemotherapy
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Drug: Systemic chemotherapy combined with immunotherapy — The electronic medical record system was used to collect patients' basic information and treatment plan information, including treatment plan, administration cycle, administration date, administration dose, frequency, number of cycles, efficacy, adverse reactions, etc.

SUMMARY:
This study focused on the longitudinal tumor burden profile (tumor macro features, histopathological types and imaging features, etc.), liver function, health status, tumor biomarkers, and serological indicators of patients with unresectable biliary malignancies before chemotherapy combined with immunotherapy to build a dynamic prediction model. Based on this model, risk stratification of BTC patients was realized to explore which specific populations could safely initiate combination therapy. By constructing a risk stratification model, it can help clinicians to screen the best treatment population and provide a basis for safe treatment of high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Confirmed by histopathological diagnosis and/or clinical diagnosis (typical imaging features, clinical manifestations, laboratory examination, etc.) as biliary malignancy (Chinese Society of Clinical Oncology (CSCO) Guidelines for Diagnosis and Treatment of Biliary malignancy (2024)); 2. Based on unresectable malignant tumor in the diagnosis of biliary and in patients undergoing chemotherapy with immunosuppressant therapy system; 3. The liver function class for Child - Pugh, A or B; 4. More than 18 years of age, gender not limited; 5. Expected survival time for 3 months or more; 6. ECOG PS score 2 or less; 7. Meet the following laboratory test parameters:

  1. Hematological system function: Absolute neutrophil count ≥ 1.0×10⁹/L; platelet count ≥ 50×10⁹/L; hemoglobin ≥ 90 g/L; international normalized ratio less than 1.7 or prothrombin time prolongation not exceeding 4 seconds.
  2. Liver function: Alanine aminotransferase/aspartate aminotransferase not exceeding 5 times the upper limit of normal; total bilirubin ≤ 210 μmol/L [≤ 2.38 mg/dL]; albumin ≥ 28 g/L.
  3. Renal function: Serum creatinine not exceeding 1.5 times the upper limit of normal.

Exclusion Criteria:

* Malignant tumors other than BTC;
* Moderate to severe ascites (ascites reaching a Child-Pugh score of 3);
* Any local treatment (including transcatheter interventional therapy, ablation therapy, internal/external radiotherapy, etc.) or surgical resection or traditional Chinese medicine within 4 weeks before the combination of systemic chemotherapy and immunotherapy;
* Incomplete data, such as incomplete laboratory test data, missing or poor-quality imaging data, or lack of prognostic information;
* Severe liver dysfunction, such as decompensated cirrhosis and other liver diseases that significantly affect bilirubin levels;
* Severe comorbidities, such as refractory hypertension (blood pressure still higher than 150/100 mm Hg after optimal drug treatment), persistent arrhythmia (CTCAE grade 2 or above), any degree of atrial fibrillation, prolonged QTc interval (more than 450 milliseconds in men and more than 470 milliseconds in women), renal insufficiency, etc.;
* Human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome;
* Pregnant or lactating women;
* Acute or chronic mental disorders (including mental disorders that affect the subject's enrollment, treatment intervention, and follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of this project is patients diagnosed with unresectable biliary malignancies and treated with systemic chemotherapy combined with immunosuppressive agents.
Sampling Method: Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1, modified Response Evaluation Criteria in Solid Tumors and immune-modified Response Evaluation Criteria In Solid Tumors(RECIST 1.1, mRECIST and iRECIST) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST 1.1, mRECIST and iRECIST) or death due to any cause, whichever occurs first.
Objective response rate(ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1, modified Response Evaluation Criteria in Solid Tumors and immune-modified Response Evaluation Criteria In Solid Tumors(RECIST 1.1, mRECIST and iRECIST) | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1, mRECIST and iRECIST.
Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors Version 1.1, modified Response Evaluation Criteria in Solid Tumors and immune-modified Response Evaluation Criteria In Solid Tumors(RECIST 1.1, mRECIST and iRECIST) | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD)per RECIST 1.1, mRECIST and iRECIST.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (2):
- China (2):
  - Zhongda Hospital,, Nanjing, Jiangsu
  - Zhongda Hospital, Nanjing, Jiangsu